CLINICAL TRIAL: NCT01411475
Title: Classification of Bifurcation Restenosis: a Prognostic Assessment
Brief Title: Prognostic Assessment of Different Pattern of Bifurcation Restenosis
Acronym: LATINA
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues
Sponsor: Ospedale Santa Maria Goretti (Other)
Responsible Party: Principal Investigator, Gregory Sgueglia, MD, Principal investigator, Ospedale Santa Maria Goretti
Other Study IDs: SMG-009
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: In-stent Coronary Artery Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bifurcation restenosis: Patients with either a main vessel or a side branch restenosis following succesful percutaneous coronary intervention
  Interventions: Other: Bifurcation restenosis classification

INTERVENTIONS:
Other: Bifurcation restenosis classification — Classification of restenosis involving coronary bifurcation according to their pattern

SUMMARY:
The LATINA registry aims at assessing a new classification of bifurcation restenosis in the prediction of major adverse cardiac events in patients who have previously undergone a succesful percutaneous bifurcation intervention.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* restenosis involving a coronary bifurcation previously treated percutaneously

Exclusion Criteria:

* life expectancy >1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 12 months
  Number of patients experiencing any of the following events: cardiac death, non-fatal miocardial infarction, target vessel revascularization

SECONDARY OUTCOMES:
Cardiac death | 12
  Number of patients experiencing a cardiac death event
Non-fatal myocardial infarction | 12 months
  Number of patients experiencing a non-fatal myocardial infarction event
Target vessel revascularization | 12 month
  Number of patients experiencing a target vessel revascularization event

CONTACTS AND LOCATIONS:
Locations (1):
- S.M. Goretti, Latina, Italy

REFERENCES:
- [Background] Sgueglia GA, Todaro D, Stipo A, Pucci E. Simultaneous inflation of two drug-eluting balloons for the treatment of coronary bifurcation restenosis: a concept series. J Invasive Cardiol. 2011 Nov;23(11):474-6. PMID 22045082